CLINICAL TRIAL: NCT04792619
Title: The Effect of Scapular Exercises on Trunk Control in Patients With Stroke: A Double-blind Randomized Study
Brief Title: The Effect of Scapular Exercises in Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Mehmet Duray, Principal Investigator, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 60116787-020/81392
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental)
  Interventions: Other: Bobath Approach
- Study (Active Comparator)
  Interventions: Other: Bobath Approach; Other: Isometric scapular exercises

INTERVENTIONS:
Other: Bobath Approach — The patients in both groups were treated with the exercise program according to the Bobath concept was planned taking the functional needs of the survivors into account, including stretching and facilitation of latissimus dorsi muscle, facilitation of abdominal muscles, placing exercises, training of lumbar spine stabilizers, functional reach of shoulder in different directions. Five sessions of about an hour each were provided to the patients
Other: Isometric scapular exercises — Isometric scapular exercises were performed to the patients included to the study group in a sitting position and at 900 of the shoulder flexion and 900 of the shoulder abduction. The patients were exercised by a physiotherapist using isometric contraction in protraction and retraction by a physiotherapist. Isometric contractions lasted 5 seconds and each exercise was repeated 2x15 times. One minute rest period was given between sets
  Arms: Study

SUMMARY:
There is a paucity of research on the correlation between postural control and upper extremity function. Analyzing the mechanisms of postural deficits and related problems is believed to give idea for any conceivable advance in future rehabilitation strategies in patients with stroke.

The purpose of this study was to examine the effect of scapular exercises on the scapular stability and trunk control. We hypothesized that scapular exercises correct the scapular position and improve postural control. Hence the reaching out movement can be applied in a controlled and fluent manner at the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed as acute stroke, being able to sit without support, presence of hemiparesis, clinical stability

Exclusion Criteria:

Shoulder joint dysfunction due to previous musculoskeletal disease, severe dementia, severe visual disturbances that could not be corrected with glasses, severe aphasia, scored ≥ 3 on the Modified Ashworth Scale and refused to participate

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Scapular mobility | 12 months
  Distance between medial border of scapula and columna vertebralis
Trunk Impairment Scale | 12 months
  postural control ability of the trunk
Trunk Control Test | 12 months
  Trunk Control
Modified Barthel Index | 12 months
  evaluate the level of disability during daily life activities
Reaching Performance Test | 12 months
  Reaching Performance

CONTACTS AND LOCATIONS:
Locations (1):
- Mehmet Duray, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No